CLINICAL TRIAL: NCT05573997
Title: Clinical Value of Novel Echocardiographic Biomarkers Assessing the Myocardial Work in Heart Failure
Brief Title: Novel Echocardiographic Biomarkers Assessing the Myocardial Work in Heart Failure
Acronym: Beyond-MyoHF
Status: Recruiting | Type: Observational
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Sponsor
Other Study IDs: 19/2022
Record Dates: First submitted 2022-10-02; First posted 2022-10-10 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Cardiovascular Diseases; Heart Failure; Valvular Heart Disease; Biochemical Dysfunction
Keywords: Heart Failure; Echocardiography; Myocardial Work; Functional Valvular Heart Disease
MeSH Terms: conditions — Cardiovascular Diseases; Heart Failure; Heart Valve Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Heart failure with reduced ejection fraction: Left Ventricular Ejection Fraction of ≤40%
  Interventions: Diagnostic Test: Investigation of clinical profile, laboratory and novel echocardiographic imaging biomarkers
- Heart failure with mid-range ejection fraction: Left Ventricular Ejection Fraction of 41-49%
  Interventions: Diagnostic Test: Investigation of clinical profile, laboratory and novel echocardiographic imaging biomarkers
- Heart failure with preserved ejection fraction: Left Ventricular Ejection Fraction of ≥50%
  Interventions: Diagnostic Test: Investigation of clinical profile, laboratory and novel echocardiographic imaging biomarkers

INTERVENTIONS:
Diagnostic Test: Investigation of clinical profile, laboratory and novel echocardiographic imaging biomarkers — Complete and comprehensive medical interview will be conducted in each eligible patient. In addition, patient's laboratory data will be recorded on admission and pre-discharge. Each patient will undergo a full echocardiographic examination with a specific protocol upon admission and pre-discharge. This will include among others 2-dimensional speckle-tracking analysis of all cardiac chambers, and non-invasive calculation of myocardial work indices of the left and right ventricle.

SUMMARY:
This study seeks to investigate the clinical value of novel echocardiographic indices, including myocardial work parameters, during the acute phase of heart failure hospitalization. The trajectory of novel echocardiographic indices from the start to the end of hospitalization will be captured, as a means to unravel and subsequently better understand the diverse pathophysiology of different phenotypes of the heart failure continuum. Correlation between novel echocardiographic indices with clinical data, biochemical data, different heart failure phenotypes, and therapeutic maneuvers will be attempted. Prognostic implications of those indices will be explored.

DETAILED DESCRIPTION:
Despite ongoing advances in early diagnosis and therapy, heart failure (HF) represents a worldwide health burden with high in-hospital mortality during the acute phase of hospitalization and high readmission rates following the event of decompensation. Patients acutely hospitalized for HF represent a widely heterogenous population in terms of primary etiology, clinical manifestations, echocardiographic characteristics, appropriate therapeutic management, and prognosis.

As more advanced HF therapeutic strategies are emerging, the cardiology community attempts to identify new HF sub-phenotypes that will serve as successful recipients of such treatments. The role of echocardiography in this attempt is far from exhausted, as novel indices are entering the research arena potentially capable of identifying new phenotypes, enlightening the subtending pathophysiology, and providing incremental prognostic information.

All adult patients acutely admitted at the Department of Cardiology at AHEPA University General Hospital of Thessaloniki with symptoms and/or signs of HF meeting the inclusion criteria will be invited to participate in the present study. A complete and comprehensive medical interview will be conducted in each eligible patient. Demographic characteristics and baseline medical history, including primary etiology and clinical presentation of hospitalization will be recorded for all participants. Pharmacological and non-pharmacological standard of care therapeutic maneuvers during the acute phase of hospitalization, as well as medical therapy upon admission and discharge will be collected. A comprehensive transthoracic echocardiographic assessment (TTE) including 2-dimensional-speckle-tracking analysis of all cardiac chambers, and non-invasive calculation of myocardial work of the left and right ventricle will be performed during hospitalization. The first TTE will be performed within 24 hours from admission, and the second within 24 hours pre-discharge, to capture the trajectory and net variations of all echocardiographic indices of interest. Blood samples for biochemical analysis, including N-terminal pro-B-type natriuretic peptide plasma concentrations will be collected upon admission and prior to discharge.

Through this prospective registry, association of novel echocardiographic indices and their net changes during hospitalization with clinical and biochemical data, diverse HF phenotypes, therapeutic maneuvers, and response to treatment will be attempted, as a means to explore the pathophysiology of different HF phenotypes and ultimately provide individualized acute HF management guidance. The clinical value and prognostic implications of those echocardiographic indices will be investigated during follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Patients acutely admitted at the Department of Cardiology of AHEPA University General Hospital, Thessaloniki, Greece with symptoms and/or signs of heart failure (HF), as those are defined by the European Society of Cardiology.
2. Patients with abnormal plasma concentration of N-terminal pro-B-type natriuretic peptide, measured within 24 hours from admission
3. Objective echocardiographic evidence of cardiac structural and/or functional abnormalities consistent with the presence of left ventricular (LV) systolic dysfunction/diastolic dysfunction/raised LV filling pressures upon admission assessment

Exclusion Criteria:

1. Symptoms and/or signs of HF secondary to congenital heart disease, infective endocarditis, pericardial disease, and history of recent cardiac surgery (<1 month)
2. Patients receiving maintenance hemodialysis
3. Patients with active malignancy and/or life expectancy < 1 year
4. Poor echocardiographic acoustic windows precluding reliable assessment and/or analysis
5. Heart transplantation
6. Patients not providing informed written consent to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients acutely admitted at the Department of Cardiology of AHEPA University General Hospital, Thessaloniki, Greece with symptoms and/or signs of heart failure, as those are specified by most updated guidelines, will be considered for enrollment in the present study. All participants will have elevated plasma concentration of N-terminal pro-B-type natriuretic peptide, measured within 24 hours from admission as well as objective echocardiographic evidence of cardiac structural and/or functional abnormalities consistent with the presence of left ventricular (LV) systolic dysfunction/diastolic dysfunction/raised LV filling pressures upon admission assessment.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-04-10 (Actual); Primary Completion 2024-12-10 (Estimated); Study Completion 2025-01-10 (Estimated)

PRIMARY OUTCOMES:
Relationship between different heart failure sub-groups and echocardiographic indices | 12 months
  Conventional and novel echocardiographic parameters including among others left ventricular myocardial work indices, right ventricular myocardial work indices, 2-dimensional speckle-tracking analysis of all cardiac chambers.

SECONDARY OUTCOMES:
Relationship between therapeutic management of acute heart failure, laboratory profile, and net changes of echocardiographic indices | 12 months
  Pharmacological and non-pharmacological therapeutic management of acute heart failure, duration of hospitalization, and laboratory profile with net variations of conventional and novel echocardiographic parameters including among others left ventricular myocardial work indices, right ventricular myocardial work indices, and 2-dimensional speckle-tracking analysis of all cardiac chambers.
Prognostic factors in acute and chronic heart failure | 12 months
  Clinical, laboratory, and echocardiographic parameters including among others left ventricular myocardial work indices, right ventricular myocardial work indices, 2-dimensional speckle-tracking analysis of all cardiac chambers.
  Different units of measure in this outcome do not represent different outcome measures. All clinical, laboratory and echocardiographic measurements will be evaluated separately in their own unit of measurement to assess potential prognostic biomarkers in patients with heart failure. This does not render the measurement of each parameter a different clinical outcome.
Relationship between clinical, laboratory, and echocardiographic biomarkers with short- and long-term prognosis of patients | 12 months
  Clinical, laboratory, and echocardiographic parameters including among others left ventricular myocardial work indices, right ventricular myocardial work indices, 2-dimensional speckle-tracking analysis of all cardiac chambers.

CONTACTS AND LOCATIONS:
Overall Officials: Vasileios Kamperidis, MD, MSc, PhD, Study Director — School of Medicine, Aristotle University of Thessaloniki; Antonios Ziakas, MD, PhD, Study Chair — Information provided by (Responsible Party):
Locations (1):
- AHEPA University Hospital, Thessaloniki, Greece, Thessaloniki, Central Macedonia, Greece

REFERENCES:
- [Derived] Anastasiou V, Stavropoulou E, Peteinidou E, Nikolaidou A, Daios S, Fardoulis E, Karamitsos T, Giannakoulas G, Naka KKappa, Delgado V, Ziakas A, Kamperidis V. Dynamic Changes in Right Ventricular-Pulmonary Arterial Coupling During Acute Heart Failure Hospitalization: Prognostic Implications. Am J Cardiol. 2025 Dec 28;262:6-15. doi: 10.1016/j.amjcard.2025.12.010. Online ahead of print. PMID 41468984
- [Derived] Anastasiou V, Papazoglou AS, Daios S, Peteinidou E, Nikolaidou A, Fardoulis E, Didagelos M, Karamitsos T, Giannakoulas G, Delgado V, Ziakas A, Kamperidis V. Prognostic Role of Right Atrial Reservoir Strain in Acute Heart Failure. Can J Cardiol. 2025 Oct;41(10):2085-2095. doi: 10.1016/j.cjca.2025.06.010. Epub 2025 Jun 23. PMID 40562231